CLINICAL TRIAL: NCT01298739
Title: Asthma Control Study 2011
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RHU-XXX-2011/1
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Asthma Control Level
Keywords: asthma control level , ACQ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Asthma control study 2011

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic patients above 18 y

Exclusion Criteria:

* COPD
* pulmonary cancer
* pulmonary tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients above 18 y
Sampling Method: Non-Probability Sample
Enrollment: 1524 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Asthma control level | 2 times

SECONDARY OUTCOMES:
Routine Therapeutical habits in control maintenance | 2 time

CONTACTS AND LOCATIONS:
Overall Officials: György Losonczy, MD PHD, Principal Investigator — Semmelweis University Budapest Pulmonology Clinic
Locations (53):
- Hungary (53):
  - Research Site, Adásztevel, Adásztevel
  - Research Site, Ajka, Ajka
  - Research Site, Albertirsa, Albertirsa
  - Research Site, Baja, Baja
  - Research Site, Balatonendréd, Balatonendréd
  - Research Site, Békés, Bekes County
  - Research Site, Budajenő, Budajenő
  - Research Site, Budakeszi, Budakeszi
  - Research Site, Budapest, Budapest
  - Research Site, Békéscsaba, Békéscsaba
  - Research Site, Celldömölk, Celldömölk
  - Research Site, Dabas, Dabas
  - Research Site, Debrecen, Debrecen
  - Research Site, Dombóvár, Dombóvár
  - Research Site, Dunaújváros, Dunaújváros
  - Research Site, Edelény, Edelény
  - Research Site, Eger, Eger
  - Research Site, Encs, Encs
  - Research Site, Esztergom, Esztergom
  - Research Site, Gyula, Gyula
  - Research Site, Gyöngyös, Gyöngyös
  - Research Site, Győr, Győr
  - Research Site, Hatvan, Hatvan
  - Research Site, Hódmezővásárhely, Hódmezővásárhely
  - Research Site, Kaposvár, Kaposvár
  - Research Site, Kecskemét, Kecskemét
  - Research Site, Kisbér, Kisbér
  - Research Site, Kiskunfélegyháza, Kiskunfélegyháza
  - Research Site, Kiskunhalas, Kiskunhalas
  - Research Site, Komárom, Komárom
  - Research Site, Körmend, Körmend
  - Research Site, Lenti, Lenti
  - Research Site, Miskolc, Miskolc
  - Research Site, Monor, Monor
  - Research Site, Mosdós, Mosdós
  - Research Site, Mátraháza, Mátraháza
  - Research Site, Mór, Mór
  - Research Site, Nagykanizsa, Nagykanizsa
  - Research Site, Nyíregyháza, Nyíregyháza
  - Research Site, Paks, Paks
  - Research Site, Pécs, Pécs
  - Research Site, Sopron, Sopron
  - Research Site, Szarvas, Szarvas
  - Research Site, Szeged, Szeged
  - Research Site, Szombathely, Szombathely
  - Research Site, Székesfehérvár, Székesfehérvár
  - Research Site, Tatabánya, Tatabánya
  - Research Site, Tata, Tata
  - Research Site, Tiszaújváros, Tiszaújváros
  - Research Site, Törökbálint, Törökbálint
  - Research Site, Törökszentmiklós, Törökszentmiklós
  - Research Site, Veszprém, Veszprém megye
  - Research Site, Zalaegerszeg, Zalaegerszeg